CLINICAL TRIAL: NCT05224856
Title: A Phase 3, Randomized, Parallel-group, Placebo-controlled, Double-blind Study to Evaluate the Efficacy and Safety of Inhaled CT-P63 and CT-P66 Combination Therapy in Symptomatic Patients With Coronavirus Disease 2019 (COVID-19) Not Requiring Supplemental Oxygen
Brief Title: To Evaluate the Safety and Efficacy of Inhaled CT-P63 and CT-P66 Combination Therapy in Symptomatic Patients With COVID-19 Not Requiring Supplemental Oxygen
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The sponsor has decided to stop development of the inhaled CT-P63/66 combination therapy.
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P63/66 3.1
Record Dates: First submitted 2022-02-03; First posted 2022-02-04 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — CT-P63; CT-P66

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-P63 and CT-P66 (Experimental)
  Interventions: Biological: CT-P63 and CT-P66 / Placebo
- Placebo (Placebo Comparator)
  Interventions: Biological: CT-P63 and CT-P66 / Placebo

INTERVENTIONS:
Biological: CT-P63 and CT-P66 / Placebo — Inhalation

SUMMARY:
This is a Phase 3 study to assess the efficacy about therapeutic effect of inhaled CT-P63 and CT-P66 combination therapy to symptomatic patiemts with COVID-19 and overall safety.

DETAILED DESCRIPTION:
CT-P63 and CT-P66 are monoclonal antibodies targeted against SARS-CoV-2 spike receptor binding domain as a treatment for COVID-19 infection. CT-P63 and CT-P66 are currently being developed by the Sponsor as a potential treatment for COVID-19 infection. In this study, efficacy, safety, and virology of inhaled CT-P63 and CT-P66 will be evaluated in symptomatic patients with COVID-19 Infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patient, aged 18 or above.
* Patient diagnosed with SARS-CoV-2 infection at Screening by using the sponsor-supplied rapid SARS-CoV-2 diagnostic test or RT-PCR.
* Patient with conditions meeting all of the following criteria:

  1. Oxygen saturation ≥ 94% on room air.
  2. Not requiring supplemental oxygen.
* Patient who has onset of one or more of the SARS-CoV-2 infection associated symptoms within 7 days prior to the study drug administration.

Exclusion Criteria:

* Patient with current serious condition meeting one of the following:

  1. Previously or currently hospitalized or requires hospitalization for treatment of serious SARS-CoV-2 related conditions.
  2. Respiratory distress with respiratory rate ≥30 breaths/min.
  3. Severe pneumonia
  4. Requires supplemental oxygen
  5. Experience shock
  6. Complicated with other organs failure, and intensive care unit monitoring treatment is needed by investigator's discretion.
* Patient who has received or has a plan to receive any of following prohibited medications or treatments:

  1. Drugs with actual or possible antiviral drugs and/or possible anti-SARS-CoV-2 activity including but not limited to nirmatrelvir and ritonavir, molnupiravir, remdesivir, chloroquine, hydroxychloroquine, dexamethasone (or alternative corticosteroids to dexamethasone), and other immunomodulatory agents and human immunodeficiency virus protease inhibitors for therapeutic purpose of SARS-CoV-2 infection prior to study drug administration
  2. Any SARS-CoV-2 human intravenous immunoglobulin, convalescent plasma for the treatment of COVID-19 infection prior to study drug administration
  3. Any approved monoclonal antibody (sotrovimab, casirivimab and imdevimab, bamlanivimab and etesevimab, etc), any other investigational device or medical product including but not limited to any monoclonal antibody(tocilizumab, sarilumab, etc.), fusion proteins or biologics for the treatment of COVID-19 infection prior to the first study drug administration.
  4. Any investigational vaccine for SARS-CoV-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Time to clinical recovery | Up to Day 14
  To evaluate the therapeutic efficacy of CT-P63 and CT-P66 combination therapy as of clinical recovery of the patients' COVID-19 symptoms.

SECONDARY OUTCOMES:
Overall safety | Up to Day 90
  To evaluate overall safety of inhaled CT-P63 and CT-P66

IPD SHARING:
Plan to Share IPD: No